CLINICAL TRIAL: NCT01021904
Title: Primary and Secondary Prevention of Human Papillomavirus (HPV) Disease in China
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: You-Lin Qiao, M.D, Ph.D. Professor and Chief, Dept of Cancer Epidemiology, Cancer Hospital/Institute, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 37207
Record Dates: First submitted 2009-11-27; First posted 2009-11-30 (Estimated); Last update posted 2009-11-30 (Estimated); Status verified 2009-11

CONDITIONS: HPV Infections; Precancerous Disease of the Cervix; Cervical Cancer; HPV Related Diseases
Keywords: Primary prevention; HPV Vaccination; HPV Infection; Cervical Cancer; HPV Related Diseases
MeSH Terms: conditions — Papillomavirus Infections; Uterine Cervical Neoplasms | interventions — Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: Gardasil (VLP, HPV Quadrivalent prophylactic vaccine) — 0.5cc I/M Site deltoid Lt Rt 3-dose regimen: 0, 2, 6 months

SUMMARY:
In a hospital-based multi-center study in China, HPV 16 was found to be the predominant type (72.9%) in cervical cancer, followed by HPV 18(8.0%) which indicated that if the HPV prophylactic vaccine are wisely applied in China, about 80% of cervical cancer can be prevented.The reported prevalence of HPV in the female population in China was about 13.2%, with women in the study between ages 15-55. HPV prevalence peaks in young adults (ages 20-24:15.5%) and pre-menopausal women (ages 45-49:15%) and this suggests an underestimation of cervical cancer burden in China.

So far, there is no nation wide organized screening program in China, nor is the vaccine available for girls innocent to HPV infection. This study aims to vaccinate the daughters (aged between 13-15 yrs) living in the selected study areas thus to evaluate how cervical cancer and other HPV related diseases can be curbed through primary and secondary prevention(in company to screening the mothers aged 35-54 yrs) and to develop a China specific model for cervical cancer prevention through HPV vaccination and HPV DNA test (careHPV).

DETAILED DESCRIPTION:
Selection of Vaccination age group

-It is well acknowledged that preadolescent or adolescent girls before their sexual debut will benefit the most from HPV vaccination. According to our previous study conducted in year 2007, the median age of sexual debut in Xinjiang was 17 years old (95% CI: 14-21). Data on the age of sexual debut in the other two identified regions is not available and we made an approximate estimation according to our data previously collected from other parts of China.From these data, we don't see an obvious time trend of sexual debut age from other parts of China and the majority of girls became sexually active after 15 years old. We thus suggest coverage of 13-15 years old girls for HPV vaccination in our identified regions.

Goal of this Program

-The purpose of this program is to implement and evaluate what it takes to establish and operate a public health program on cervical cancer prevention by vaccination and early detection treatment program in resource restricted selected autonomous regions of China. The learnings on how to implement such projects and the costing of the interventions and program will be useful for national policy planners and regional authorities when they consider future health priorities and allocation of resources.

Objectives

The objectives of the pilot program are to:

1. Develop a communication and education program on cervical cancer for families in the target area and try to deliver the message of 'Vaccinate the daughters and screen the mothers' to curb cervical cancer.
2. Develop a China specific model for cervical cancer prevention through HPV vaccination and HPV DNA test ( careHPV).
3. Capacitate the health facilities in the selected counties in each region to conduct HPV vaccination, screen for cervical cancer and treat precancerous lesions and cervical cancer.
4. Develop a referral system for advanced cases of cervical cancer that cannot be treated at lower level facilities
5. Develop training guidelines and supportive management systems for all levels of the health care system and cost all interventions for policy purposes.

ELIGIBILITY:
Inclusion Criteria:

* Long term residence in the selected study areas (at least more than 5 years from the beginning of the study)
* aged between 13-15 yrs
* With complete cervix
* Not sexually active
* Physically competent to undergo vaccination
* With ability to provide informed consent

Exclusion Criteria:

* Short term residence (less than 5 years from the beginning of the study)
* Dose not have a cervix
* Physically incompetent to undergo vaccination
* With no ability to provide informed consent

Ages: 13 Years to 15 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 6200 (Estimated)
Dates: Start 2010-06; Primary Completion 2014-06 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
The quadrivalent HPV vaccine can prevent HPV naive girls at baseline from being infected at least on a five year follow-up and longer. | 5 years

SECONDARY OUTCOMES:
Knowledge of HPV and the link between HPV and cervical cancer | 5 years
Attitudes towards HPV vaccine | 5 years
Attitudes towards sex and the proper age of sexual debut; | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: You-lin Qiao, M.D. Ph.D., Principal Investigator — Cancer Hospital/Institute, Chinese Academy of Medical Sciences

REFERENCES:
- [Background] Munoz N. Human papillomavirus and cancer: the epidemiological evidence. J Clin Virol. 2000 Oct;19(1-2):1-5. doi: 10.1016/s1386-6532(00)00125-6. PMID 11091143
- [Background] Bosch FX, Lorincz A, Munoz N, Meijer CJ, Shah KV. The causal relation between human papillomavirus and cervical cancer. J Clin Pathol. 2002 Apr;55(4):244-65. doi: 10.1136/jcp.55.4.244. PMID 11919208
- [Background] Trottier H, Franco EL. The epidemiology of genital human papillomavirus infection. Vaccine. 2006 Mar 30;24 Suppl 1:S1-15. doi: 10.1016/j.vaccine.2005.09.054. PMID 16406226
- [Background] Schiffman M, Castle PE. Human papillomavirus: epidemiology and public health. Arch Pathol Lab Med. 2003 Aug;127(8):930-4. doi: 10.5858/2003-127-930-HPEAPH. PMID 12873163
- [Background] Franco EL, Harper DM. Vaccination against human papillomavirus infection: a new paradigm in cervical cancer control. Vaccine. 2005 Mar 18;23(17-18):2388-94. doi: 10.1016/j.vaccine.2005.01.016. PMID 15755633
- [Background] Munoz N, Bosch FX, de Sanjose S, Herrero R, Castellsague X, Shah KV, Snijders PJ, Meijer CJ; International Agency for Research on Cancer Multicenter Cervical Cancer Study Group. Epidemiologic classification of human papillomavirus types associated with cervical cancer. N Engl J Med. 2003 Feb 6;348(6):518-27. doi: 10.1056/NEJMoa021641. PMID 12571259
- [Background] Cox JT. Epidemiology and natural history of HPV. J Fam Pract. 2006 Nov;Suppl:3-9. PMID 17366752
- [Background] Padel AF, Venning VA, Evans MF, Quantrill AM, Fleming KA. Human papillomaviruses in anogenital warts in children: typing by in situ hybridisation. BMJ. 1990 Jun 9;300(6738):1491-4. doi: 10.1136/bmj.300.6738.1491. PMID 2164854
- [Background] Sugase M, Moriyama S, Matsukura T. Human papillomavirus in exophytic condylomatous lesions on different female genital regions. J Med Virol. 1991 May;34(1):1-6. doi: 10.1002/jmv.1890340102. PMID 1653304
- [Background] Qiao YL, Sellors JW, Eder PS, Bao YP, Lim JM, Zhao FH, Weigl B, Zhang WH, Peck RB, Li L, Chen F, Pan QJ, Lorincz AT. A new HPV-DNA test for cervical-cancer screening in developing regions: a cross-sectional study of clinical accuracy in rural China. Lancet Oncol. 2008 Oct;9(10):929-36. doi: 10.1016/S1470-2045(08)70210-9. Epub 2008 Sep 19. PMID 18805733